CLINICAL TRIAL: NCT06330311
Title: Effectiveness of Whole-Body Vibration on Lower Limb Motor Function and Spasticity in Children With Spastic Cerebral Palsy
Brief Title: Effectiveness of Whole-Body Vibration
Acronym: WBVibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, MARIA JOSE DIAZ ARRIBAS, Tenured Proffesor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/551-EC
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Spastic Cerebral Palsy; Physical Therapy Modalities; Vibration; Exposure; Lower Extremity Weakness, Spastic; Muscle Spasticity
Keywords: Spastic Cerebral Palsy; Physical Therapy; Whole-Body Vibration; Gross Motor Function; Lower Limb Spasticity
MeSH Terms: conditions — Cerebral Palsy; Paraparesis, Spastic; Muscle Spasticity | interventions — Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to experimental or control group
Who Masked: Investigator
Masking Description: The principal investigator will be blinded to the randomization, patient assessment, and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Body Vibration Group (Experimental): Allocated participants will receive an intervention with Whole-Body vibration (12 - 18 minutes, 12 - 20 hz, 1 - 2 mm progression) added to a physical therapy treatment based on learning and motor control through activities with a defined goal and therapeutic exercises (56 minutes per session) 4 sessions per week for 4 weeks.
  Interventions: Other: Physiotherapy
- Control Group (Active Comparator): Physical therapy treatment based on learning and motor control through activities with a defined goal and therapeutic exercises (56 minutes per session) 4 sessions per week for 4 weeks.
  In the control group, the same measurements will be made at the same time as the subjects in the experimental group.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Evidence-based multimodal physiotherapy treatment based on learning and motor control
  Other Names: Therapeutic exercise

SUMMARY:
Cerebral Palsy is the most common cause of severe physical disability in childhood and may present difficulties and limitations that will have an impact on their independence and integration in all social areas.

Within interventions aiming to manage CP Whole-Body Vibration (WBV) has shown some benefits such as reducing spasticity or improving strength and functionality of the lower limbs.

The aim of this study is to assess the effectiveness on motor function and spasticity of the lower limbs by adding an intervention with WBV to an evidence-based multimodal physiotherapy treatment in children with CP.

DETAILED DESCRIPTION:
Cerebral Palsy is the most common cause of severe physical disability in childhood (1.5 - 3 cases per thousand live births) and may or may not be accompanied by intellectual, sensory, communication deficits and epileptic syndromes depending on the brain region affected. The most frequent form of presentation is spastic cerebral palsy, characterized by atypical motor development, abnormal movement or posture, hyperreflexia, and increased muscle tone. These difficulties and limitations will have an impact on their independence and integration in all social areas.

The use of Whole-Body Vibration (WBV) to reduce spasticity of the lower limb and thereby improve functionality has been used for more than a decade showing some benefits such as reducing spasticity or improving strength and functionality of the lower limbs.

The purpose of this randomized controlled trial is to assess the effectiveness on motor function and spasticity of the lower limbs by adding an intervention with WBV to an evidence-based multimodal physiotherapy treatment in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spastic cerebral palsy.
* Aged between 8 and 14 years.
* GMFCS I, II or III: with the ability to walk independently with or without technical aids; with the ability to stand for 3 minutes independently or gripped on the stand; with the ability to understand and follow simple instructions; with the ability to tolerate clinical tests and examinations.

Exclusion Criteria:

* Participation in treatments with serial casting or botulinum toxin during the 3 months prior to the study.
* Recent orthopedic surgery (less than 12 months).
* Participation in other muscle strengthening programs during the 4 months prior to this clinical study.
* Children who have developed fixed contractures in lower limbs joints.
* Medical conditions where physical exercise is contraindicated.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
GROSS MOTOR FUNCTION MEASURE 88 (D and E dimensions) | Baseline
  GROSS MOTOR FUNCTION MEASURE 88 is a clinical test to evaluate changes in gross motor function over time in children and youth with cerebral palsy.
  The GROSS MOTOR FUNCTION MEASURE 88 is divided in 5 dimensions:
  A: Lying and rolling.
  The minimum value is 0 and the maximum value is 51. Higher scores mean better outcome.
  B: Sitting.
  The minimum value is 0 and the maximum value is 60. Higher scores mean better outcome.
  C: Crawling and Kneeling.
  The minimum value is 0 and the maximum value is 42. Higher scores mean better outcome.
  D: Standing.
  The minimum value is 0 and the maximum value is 39. Higher scores mean better outcome.
  E: Walking, running and jumping.
  The minimum value is 0 and the maximum value is 72. Higher scores mean better outcome.
  The minimum value overall of the GROSS MOTOR FUNCTION MEASURE 88 is 0 and the maximum value overall is 264. Higher scores mean better outcome.
GROSS MOTOR FUNCTION MEASURE 88 (D and E dimensions) | 1 month
  GROSS MOTOR FUNCTION MEASURE 88 is a clinical test to evaluate changes in gross motor function over time in children and youth with cerebral palsy.
  The GROSS MOTOR FUNCTION MEASURE 88 is divided in 5 dimensions:
  A: Lying and rolling.
  The minimum value is 0 and the maximum value is 51. Higher scores mean better outcome.
  B: Sitting.
  The minimum value is 0 and the maximum value is 60. Higher scores mean better outcome.
  C: Crawling and Kneeling.
  The minimum value is 0 and the maximum value is 42. Higher scores mean better outcome.
  D: Standing.
  The minimum value is 0 and the maximum value is 39. Higher scores mean better outcome.
  E: Walking, running and jumping.
  The minimum value is 0 and the maximum value is 72. Higher scores mean better outcome.
  The minimum value overall of the GROSS MOTOR FUNCTION MEASURE 88 is 0 and the maximum value overall is 264. Higher scores mean better outcome.
GROSS MOTOR FUNCTION MEASURE 88 (D and E dimensions) | 2 months
  GROSS MOTOR FUNCTION MEASURE 88 is a clinical test to evaluate changes in gross motor function over time in children and youth with cerebral palsy.
  The GROSS MOTOR FUNCTION MEASURE 88 is divided in 5 dimensions:
  A: Lying and rolling.
  The minimum value is 0 and the maximum value is 51. Higher scores mean better outcome.
  B: Sitting.
  The minimum value is 0 and the maximum value is 60. Higher scores mean better outcome.
  C: Crawling and Kneeling.
  The minimum value is 0 and the maximum value is 42. Higher scores mean better outcome.
  D: Standing.
  The minimum value is 0 and the maximum value is 39. Higher scores mean better outcome.
  E: Walking, running and jumping.
  The minimum value is 0 and the maximum value is 72. Higher scores mean better outcome.
  The minimum value overall of the GROSS MOTOR FUNCTION MEASURE 88 is 0 and the maximum value overall is 264. Higher scores mean better outcome.
GROSS MOTOR FUNCTION MEASURE 88 (D and E dimensions) | 6 months
  GROSS MOTOR FUNCTION MEASURE 88 is a clinical test to evaluate changes in gross motor function over time in children and youth with cerebral palsy.
  The GROSS MOTOR FUNCTION MEASURE 88 is divided in 5 dimensions:
  A: Lying and rolling.
  The minimum value is 0 and the maximum value is 51. Higher scores mean better outcome.
  B: Sitting.
  The minimum value is 0 and the maximum value is 60. Higher scores mean better outcome.
  C: Crawling and Kneeling.
  The minimum value is 0 and the maximum value is 42. Higher scores mean better outcome.
  D: Standing.
  The minimum value is 0 and the maximum value is 39. Higher scores mean better outcome.
  E: Walking, running and jumping.
  The minimum value is 0 and the maximum value is 72. Higher scores mean better outcome.
  The minimum value overall of the GROSS MOTOR FUNCTION MEASURE 88 is 0 and the maximum value overall is 264. Higher scores mean better outcome.
Modified Ashworth Scale (MAS) | Baseline
  The Modified Ashworth Scale is a clinical tool to measure the increase of muscle tone.
  MAS is a 6 point numerical scale that graded muscle tone from 0 to 4:
  0 = No increase in muscle tone
  1 = Slight increase in muscle tone. Minimal resistance at end of range of motion
  1+ = Slight increase in muscle tone. Minimal resistance through less than half of range of motion
  2 = More marked increase in muscle tone through most range of motion. Affected part easily moved
  3 = Considerable increase in muscle tone. Passive movement difficult
  4 = Affected part rigid in flexion or extension
Modified Ashworth Scale (MAS) | 1 month
  The Modified Ashworth Scale is a clinical tool to measure the increase of muscle tone.
  MAS is a 6 point numerical scale that graded muscle tone from 0 to 4:
  0 = No increase in muscle tone
  1 = Slight increase in muscle tone. Minimal resistance at end of range of motion
  1+ = Slight increase in muscle tone. Minimal resistance through less than half of range of motion
  2 = More marked increase in muscle tone through most range of motion. Affected part easily moved
  3 = Considerable increase in muscle tone. Passive movement difficult
  4 = Affected part rigid in flexion or extension
Modified Ashworth Scale (MAS) | 2 month
  The Modified Ashworth Scale is a clinical tool to measure the increase of muscle tone.
  MAS is a 6 point numerical scale that graded muscle tone from 0 to 4:
  0 = No increase in muscle tone
  1 = Slight increase in muscle tone. Minimal resistance at end of range of motion
  1+ = Slight increase in muscle tone. Minimal resistance through less than half of range of motion
  2 = More marked increase in muscle tone through most range of motion. Affected part easily moved
  3 = Considerable increase in muscle tone. Passive movement difficult
  4 = Affected part rigid in flexion or extension
Modified Ashworth Scale (MAS) | 6 month
  The Modified Ashworth Scale is a clinical tool to measure the increase of muscle tone.
  MAS is a 6 point numerical scale that graded muscle tone from 0 to 4:
  0 = No increase in muscle tone
  1 = Slight increase in muscle tone. Minimal resistance at end of range of motion
  1+ = Slight increase in muscle tone. Minimal resistance through less than half of range of motion
  2 = More marked increase in muscle tone through most range of motion. Affected part easily moved
  3 = Considerable increase in muscle tone. Passive movement difficult
  4 = Affected part rigid in flexion or extension

SECONDARY OUTCOMES:
6 Minute Walking Test (6MWT) | Baseline
  6MWT is a test that measures the maximum distance walked by each patient for 6 minutes, on a hard and flat 30 meters surface.
  The 6MWT assesses submaximal functional capacity. In addition to distance, the test measures oxygen saturation and heart rate.
6 Minute Walking Test (6MWT) | 1 month
  6MWT is a test that measures the maximum distance walked by each patient for 6 minutes, on a hard and flat 30 meters surface.
  The 6MWT assesses submaximal functional capacity. In addition to distance, the test measures oxygen saturation and heart rate.
6 Minute Walking Test (6MWT) | 2 month
  6MWT is a test that measures the maximum distance walked by each patient for 6 minutes, on a hard and flat 30 meters surface.
  The 6MWT assesses submaximal functional capacity. In addition to distance, the test measures oxygen saturation and heart rate.
6 Minute Walking Test (6MWT) | 6 month
  6MWT is a test that measures the maximum distance walked by each patient for 6 minutes, on a hard and flat 30 meters surface.
  The 6MWT assesses submaximal functional capacity. In addition to distance, the test measures oxygen saturation and heart rate.
Dynamometry | Baseline
  Hand dynamometer will be used to measure the strength in these muscles of the lower limbs:
  * Ankle dorsal flexion
  * Ankle plantar flexion
  * Hip flexors
  * Hip extensors
  * Knee flexors
  * Knee extensors
  * Hip abductors
Dynamometry | 1 month
  Hand dynamometer will be used to measure the strength in these muscles of the lower limbs:
  * Ankle dorsal flexion
  * Ankle plantar flexion
  * Hip flexors
  * Hip extensors
  * Knee flexors
  * Knee extensors
  * Hip abductors
Dynamometry | 2 month
  Hand dynamometer will be used to measure the strength in these muscles of the lower limbs:
  * Ankle dorsal flexion
  * Ankle plantar flexion
  * Hip flexors
  * Hip extensors
  * Knee flexors
  * Knee extensors
  * Hip abductors
Dynamometry | 6 month
  Hand dynamometer will be used to measure the strength in these muscles of the lower limbs:
  * Ankle dorsal flexion
  * Ankle plantar flexion
  * Hip flexors
  * Hip extensors
  * Knee flexors
  * Knee extensors
  * Hip abductors
Mini-Balance Evaluation System Test | Baseline
  The Mini-Balance Evaluation System Test is a balance assessment that includes 14 items in 4 categories. The 14 items are scored from 0 to 2.
  - Anticipatory
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Reactive Postural Control
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Sensory Orientation
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Dynamic Gait
  The minimum value is 0 and the maximum value is 10. Higher scores mean better outcome.
  The minimum value overall of the Mini-Balance Evaluation System is 0 and the maximum value overall is 28. Higher scores mean better outcome.
Mini-Balance Evaluation System Test | 1 month
  The Mini-Balance Evaluation System Test is a balance assessment that includes 14 items in 4 categories. The 14 items are scored from 0 to 2.
  - Anticipatory
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Reactive Postural Control
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Sensory Orientation
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Dynamic Gait
  The minimum value is 0 and the maximum value is 10. Higher scores mean better outcome.
  The minimum value overall of the Mini-Balance Evaluation System is 0 and the maximum value overall is 28. Higher scores mean better outcome.
Mini-Balance Evaluation System Test | 2 month
  The Mini-Balance Evaluation System Test is a balance assessment that includes 14 items in 4 categories. The 14 items are scored from 0 to 2.
  - Anticipatory
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Reactive Postural Control
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Sensory Orientation
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Dynamic Gait
  The minimum value is 0 and the maximum value is 10. Higher scores mean better outcome.
  The minimum value overall of the Mini-Balance Evaluation System is 0 and the maximum value overall is 28. Higher scores mean better outcome.
Mini-Balance Evaluation System Test | 6 month
  The Mini-Balance Evaluation System Test is a balance assessment that includes 14 items in 4 categories. The 14 items are scored from 0 to 2.
  - Anticipatory
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Reactive Postural Control
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Sensory Orientation
  The minimum value is 0 and the maximum value is 6. Higher scores mean better outcome.
  - Dynamic Gait
  The minimum value is 0 and the maximum value is 10. Higher scores mean better outcome.
  The minimum value overall of the Mini-Balance Evaluation System is 0 and the maximum value overall is 28. Higher scores mean better outcome.
Cerebral Palsy Quality of Life questionnaire (CP-QOL) | Baseline
  The Cerebral Palsy Quality of Life questionnaire will be used to assess several aspects of subjective happiness and well-being of children with cerebral palsy.
  It sets up a profile of qualify of life of children with CP and understand their perception of life.
  There are two versions of the CP-QOL:
  - A primary caregiver-proxy report version.
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire primary caregiver-proxy report version is 53 and the maximum value overall is 477. Higher scores mean better outcome.
  - A self-report version for children with CP
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire self-report version for children with CP is 43 and the maximum value overall is 387. Higher scores mean better outcome.
Cerebral Palsy Quality of Life questionnaire (CP-QOL) | 2 month
  The Cerebral Palsy Quality of Life questionnaire will be used to assess several aspects of subjective happiness and well-being of children with cerebral palsy.
  It sets up a profile of qualify of life of children with CP and understand their perception of life.
  There are two versions of the CP-QOL:
  - A primary caregiver-proxy report version.
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire primary caregiver-proxy report version is 53 and the maximum value overall is 477. Higher scores mean better outcome.
  - A self-report version for children with CP
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire self-report version for children with CP is 43 and the maximum value overall is 387. Higher scores mean better outcome.
Cerebral Palsy Quality of Life questionnaire (CP-QOL) | 6 month
  The Cerebral Palsy Quality of Life questionnaire will be used to assess several aspects of subjective happiness and well-being of children with cerebral palsy.
  It sets up a profile of qualify of life of children with CP and understand their perception of life.
  There are two versions of the CP-QOL:
  - A primary caregiver-proxy report version.
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire primary caregiver-proxy report version is 53 and the maximum value overall is 477. Higher scores mean better outcome.
  - A self-report version for children with CP
  The minimum value overall of the Cerebral Palsy Quality of Life questionnaire self-report version for children with CP is 43 and the maximum value overall is 387. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: María J Díaz Arribas, PhD, Study Director — Universidad Complutense de Madrid; Ángela C Álvarez Melcón, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- María José Díaz Arribas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntyre S, Goldsmith S, Webb A, Ehlinger V, Hollung SJ, McConnell K, Arnaud C, Smithers-Sheedy H, Oskoui M, Khandaker G, Himmelmann K; Global CP Prevalence Group*. Global prevalence of cerebral palsy: A systematic analysis. Dev Med Child Neurol. 2022 Dec;64(12):1494-1506. doi: 10.1111/dmcn.15346. Epub 2022 Aug 11. PMID 35952356
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350
- [Background] Kahraman A, Seyhan K, Deger U, Kutluturk S, Mutlu A. Should botulinum toxin A injections be repeated in children with cerebral palsy? A systematic review. Dev Med Child Neurol. 2016 Sep;58(9):910-7. doi: 10.1111/dmcn.13135. Epub 2016 Apr 22. PMID 27103334
- [Background] Multani I, Manji J, Hastings-Ison T, Khot A, Graham K. Botulinum Toxin in the Management of Children with Cerebral Palsy. Paediatr Drugs. 2019 Aug;21(4):261-281. doi: 10.1007/s40272-019-00344-8. PMID 31257556
- [Background] Buizer AI, Martens BHM, Grandbois van Ravenhorst C, Schoonmade LJ, Becher JG, Vermeulen RJ. Effect of continuous intrathecal baclofen therapy in children: a systematic review. Dev Med Child Neurol. 2019 Feb;61(2):128-134. doi: 10.1111/dmcn.14005. Epub 2018 Sep 6. PMID 30187921
- [Background] Hasnat MJ, Rice JE. Intrathecal baclofen for treating spasticity in children with cerebral palsy. Cochrane Database Syst Rev. 2015 Nov 13;2015(11):CD004552. doi: 10.1002/14651858.CD004552.pub2. PMID 26563961
- [Background] Health Quality Ontario. Lumbosacral Dorsal Rhizotomy for Spastic Cerebral Palsy: A Health Technology Assessment. Ont Health Technol Assess Ser. 2017 Jul 6;17(10):1-186. eCollection 2017. PMID 28757906
- [Background] Hagglund G, Alriksson-Schmidt A, Lauge-Pedersen H, Rodby-Bousquet E, Wagner P, Westbom L. Prevention of dislocation of the hip in children with cerebral palsy: 20-year results of a population-based prevention programme. Bone Joint J. 2014 Nov;96-B(11):1546-52. doi: 10.1302/0301-620X.96B11.34385. PMID 25371472
- [Background] Novak I, Hines M, Goldsmith S, Barclay R. Clinical prognostic messages from a systematic review on cerebral palsy. Pediatrics. 2012 Nov;130(5):e1285-312. doi: 10.1542/peds.2012-0924. Epub 2012 Oct 8. PMID 23045562
- [Background] Amirmudin NA, Lavelle G, Theologis T, Thompson N, Ryan JM. Multilevel Surgery for Children With Cerebral Palsy: A Meta-analysis. Pediatrics. 2019 Apr;143(4):e20183390. doi: 10.1542/peds.2018-3390. PMID 30918016
- [Background] Lamberts RP, Burger M, du Toit J, Langerak NG. A Systematic Review of the Effects of Single-Event Multilevel Surgery on Gait Parameters in Children with Spastic Cerebral Palsy. PLoS One. 2016 Oct 18;11(10):e0164686. doi: 10.1371/journal.pone.0164686. eCollection 2016. PMID 27755599
- [Background] Tekin F, Kavlak E, Cavlak U, Altug F. Effectiveness of Neuro-Developmental Treatment (Bobath Concept) on postural control and balance in Cerebral Palsied children. J Back Musculoskelet Rehabil. 2018;31(2):397-403. doi: 10.3233/BMR-170813. PMID 29171980
- [Background] Ha SY, Sung YH. Effects of Vojta approach on diaphragm movement in children with spastic cerebral palsy. J Exerc Rehabil. 2018 Dec 27;14(6):1005-1009. doi: 10.12965/jer.1836498.249. eCollection 2018 Dec. PMID 30656162
- [Background] Hadders-Algra M, Boxum AG, Hielkema T, Hamer EG. Effect of early intervention in infants at very high risk of cerebral palsy: a systematic review. Dev Med Child Neurol. 2017 Mar;59(3):246-258. doi: 10.1111/dmcn.13331. Epub 2016 Dec 7. PMID 27925172
- [Background] Das SP, Ganesh GS. Evidence-based Approach to Physical Therapy in Cerebral Palsy. Indian J Orthop. 2019 Jan-Feb;53(1):20-34. doi: 10.4103/ortho.IJOrtho_241_17. PMID 30905979
- [Background] Chiu HC, Ada L. Effect of functional electrical stimulation on activity in children with cerebral palsy: a systematic review. Pediatr Phys Ther. 2014 Fall;26(3):283-8. doi: 10.1097/PEP.0000000000000045. PMID 24819681
- [Background] Salazar AP, Pagnussat AS, Pereira GA, Scopel G, Lukrafka JL. Neuromuscular electrical stimulation to improve gross motor function in children with cerebral palsy: a meta-analysis. Braz J Phys Ther. 2019 Sep-Oct;23(5):378-386. doi: 10.1016/j.bjpt.2019.01.006. Epub 2019 Jan 23. PMID 30712812
- [Background] Wells H, Marquez J, Wakely L. Garment Therapy does not Improve Function in Children with Cerebral Palsy: A Systematic Review. Phys Occup Ther Pediatr. 2018 Nov;38(4):395-416. doi: 10.1080/01942638.2017.1365323. Epub 2017 Sep 18. PMID 28922041
- [Background] Martins E, Cordovil R, Oliveira R, Letras S, Lourenco S, Pereira I, Ferro A, Lopes I, Silva CR, Marques M. Efficacy of suit therapy on functioning in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2016 Apr;58(4):348-60. doi: 10.1111/dmcn.12988. Epub 2015 Nov 27. PMID 26613800
- [Background] Buccino G, Arisi D, Gough P, Aprile D, Ferri C, Serotti L, Tiberti A, Fazzi E. Improving upper limb motor functions through action observation treatment: a pilot study in children with cerebral palsy. Dev Med Child Neurol. 2012 Sep;54(9):822-8. doi: 10.1111/j.1469-8749.2012.04334.x. Epub 2012 Jul 6. PMID 22765352
- [Background] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Fogassi L, Cioni G. Randomized trial of observation and execution of upper extremity actions versus action alone in children with unilateral cerebral palsy. Neurorehabil Neural Repair. 2013 Nov-Dec;27(9):808-15. doi: 10.1177/1545968313497101. Epub 2013 Jul 25. PMID 23886886
- [Background] Ferre CL, Brandao M, Surana B, Dew AP, Moreau NG, Gordon AM. Caregiver-directed home-based intensive bimanual training in young children with unilateral spastic cerebral palsy: a randomized trial. Dev Med Child Neurol. 2017 May;59(5):497-504. doi: 10.1111/dmcn.13330. Epub 2016 Nov 19. PMID 27864822
- [Background] Brandao MB, Mancini MC, Ferre CL, Figueiredo PRP, Oliveira RHS, Goncalves SC, Dias MCS, Gordon AM. Does Dosage Matter? A Pilot Study of Hand-Arm Bimanual Intensive Training (HABIT) Dose and Dosing Schedule in Children with Unilateral Cerebral Palsy. Phys Occup Ther Pediatr. 2018 Aug;38(3):227-242. doi: 10.1080/01942638.2017.1407014. Epub 2017 Dec 14. PMID 29240518
- [Background] Friel KM, Kuo HC, Fuller J, Ferre CL, Brandao M, Carmel JB, Bleyenheuft Y, Gowatsky JL, Stanford AD, Rowny SB, Luber B, Bassi B, Murphy DL, Lisanby SH, Gordon AM. Skilled Bimanual Training Drives Motor Cortex Plasticity in Children With Unilateral Cerebral Palsy. Neurorehabil Neural Repair. 2016 Oct;30(9):834-44. doi: 10.1177/1545968315625838. Epub 2016 Feb 11. PMID 26867559
- [Background] Inguaggiato E, Sgandurra G, Perazza S, Guzzetta A, Cioni G. Brain reorganization following intervention in children with congenital hemiplegia: a systematic review. Neural Plast. 2013;2013:356275. doi: 10.1155/2013/356275. Epub 2013 Dec 3. PMID 24367726
- [Background] Hoare BJ, Wallen MA, Thorley MN, Jackman ML, Carey LM, Imms C. Constraint-induced movement therapy in children with unilateral cerebral palsy. Cochrane Database Syst Rev. 2019 Apr 1;4(4):CD004149. doi: 10.1002/14651858.CD004149.pub3. PMID 30932166
- [Background] Sakzewski L, Ziviani J, Boyd RN. Efficacy of upper limb therapies for unilateral cerebral palsy: a meta-analysis. Pediatrics. 2014 Jan;133(1):e175-204. doi: 10.1542/peds.2013-0675. Epub 2013 Dec 23. PMID 24366991
- [Background] Chen YP, Pope S, Tyler D, Warren GL. Effectiveness of constraint-induced movement therapy on upper-extremity function in children with cerebral palsy: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2014 Oct;28(10):939-53. doi: 10.1177/0269215514544982. Epub 2014 Aug 14. PMID 25125440
- [Background] Jamali AR, Amini M. The Effects of Constraint-Induced Movement Therapy on Functions of Cerebral Palsy Children. Iran J Child Neurol. 2018 Fall;12(4):16-27. PMID 30279705
- [Background] Fonseca PRJ, Filoni E, Melo Setter C, Marques Berbel A, Olival Fernandes A, Calhes de Franco Moura R. Constraint-induced movement therapy of upper limb of children with cerebral palsy in clinical practice: systematic review of the literature. Fisioterapia e Pesquisa. 2017;24(3):334-46.
- [Background] Chiu HC, Ada L. Constraint-induced movement therapy improves upper limb activity and participation in hemiplegic cerebral palsy: a systematic review. J Physiother. 2016 Jul;62(3):130-7. doi: 10.1016/j.jphys.2016.05.013. Epub 2016 Jun 17. PMID 27323932
- [Background] Toovey R, Bernie C, Harvey AR, McGinley JL, Spittle AJ. Task-specific gross motor skills training for ambulant school-aged children with cerebral palsy: a systematic review. BMJ Paediatr Open. 2017 Aug 11;1(1):e000078. doi: 10.1136/bmjpo-2017-000078. eCollection 2017. PMID 29637118
- [Background] Novak I, Berry J. Home program intervention effectiveness evidence. Phys Occup Ther Pediatr. 2014 Nov;34(4):384-9. doi: 10.3109/01942638.2014.964020. Epub 2014 Oct 15. No abstract available. PMID 25317927
- [Background] Booth ATC, Buizer AI, Meyns P, Oude Lansink ILB, Steenbrink F, van der Krogt MM. The efficacy of functional gait training in children and young adults with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2018 Sep;60(9):866-883. doi: 10.1111/dmcn.13708. Epub 2018 Mar 7. PMID 29512110
- [Background] Moreau NG, Bodkin AW, Bjornson K, Hobbs A, Soileau M, Lahasky K. Effectiveness of Rehabilitation Interventions to Improve Gait Speed in Children With Cerebral Palsy: Systematic Review and Meta-analysis. Phys Ther. 2016 Dec;96(12):1938-1954. doi: 10.2522/ptj.20150401. Epub 2016 Jun 16. PMID 27313240
- [Background] Lefmann S, Russo R, Hillier S. The effectiveness of robotic-assisted gait training for paediatric gait disorders: systematic review. J Neuroeng Rehabil. 2017 Jan 5;14(1):1. doi: 10.1186/s12984-016-0214-x. PMID 28057016
- [Background] Morgan C, Novak I, Badawi N. Enriched environments and motor outcomes in cerebral palsy: systematic review and meta-analysis. Pediatrics. 2013 Sep;132(3):e735-46. doi: 10.1542/peds.2012-3985. Epub 2013 Aug 19. PMID 23958771
- [Background] Kruijsen-Terpstra AJA, Ketelaar M, Verschuren O, Gorter JW, Vos RC, Verheijden J, Jongmans MJ, Visser-Meily A. Efficacy of three therapy approaches in preschool children with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2016 Jul;58(7):758-766. doi: 10.1111/dmcn.12966. Epub 2015 Nov 24. PMID 26880083
- [Background] Kleim JA, Jones TA. Principles of experience-dependent neural plasticity: implications for rehabilitation after brain damage. J Speech Lang Hear Res. 2008 Feb;51(1):S225-39. doi: 10.1044/1092-4388(2008/018). PMID 18230848
- [Background] O'Brien TD, Noyes J, Spencer LH, Kubis HP, Hastings RP, Whitaker R. Systematic review of physical activity and exercise interventions to improve health, fitness and well-being of children and young people who use wheelchairs. BMJ Open Sport Exerc Med. 2016 Nov 15;2(1):e000109. doi: 10.1136/bmjsem-2016-000109. eCollection 2016. PMID 27900176
- [Background] Reedman S, Boyd RN, Sakzewski L. The efficacy of interventions to increase physical activity participation of children with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2017 Oct;59(10):1011-1018. doi: 10.1111/dmcn.13413. Epub 2017 Mar 20. PMID 28318009
- [Background] Bloemen M, Van Wely L, Mollema J, Dallmeijer A, de Groot J. Evidence for increasing physical activity in children with physical disabilities: a systematic review. Dev Med Child Neurol. 2017 Oct;59(10):1004-1010. doi: 10.1111/dmcn.13422. Epub 2017 Apr 4. PMID 28374442
- [Background] Verschuren O, Darrah J, Novak I, Ketelaar M, Wiart L. Health-enhancing physical activity in children with cerebral palsy: more of the same is not enough. Phys Ther. 2014 Feb;94(2):297-305. doi: 10.2522/ptj.20130214. Epub 2013 Oct 3. PMID 24092902
- [Background] Gannotti ME. Coupling Timing of Interventions With Dose to Optimize Plasticity and Participation in Pediatric Neurologic Populations. Pediatr Phys Ther. 2017 Jul;29 Suppl 3(Suppl 3 IV STEP 2016 CONFERENCE PROCEEDINGS ):S37-S47. doi: 10.1097/PEP.0000000000000383. PMID 28654476
- [Background] van Vulpen LF, de Groot S, Rameckers EAA, Becher JG, Dallmeijer AJ. Effectiveness of Functional Power Training on Walking Ability in Young Children With Cerebral Palsy: Study Protocol of a Double-Baseline Trial. Pediatr Phys Ther. 2017 Jul;29(3):275-282. doi: 10.1097/PEP.0000000000000424. PMID 28654503
- [Background] Ko J, Kim M. Reliability and responsiveness of the gross motor function measure-88 in children with cerebral palsy. Phys Ther. 2013 Mar;93(3):393-400. doi: 10.2522/ptj.20110374. Epub 2012 Nov 8. PMID 23139425
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Background] Maher CA, Williams MT, Olds TS. The six-minute walk test for children with cerebral palsy. Int J Rehabil Res. 2008 Jun;31(2):185-8. doi: 10.1097/MRR.0b013e32830150f9. PMID 18467936
- [Background] Nsenga Leunkeu A, Shephard RJ, Ahmaidi S. Six-minute walk test in children with cerebral palsy gross motor function classification system levels I and II: reproducibility, validity, and training effects. Arch Phys Med Rehabil. 2012 Dec;93(12):2333-9. doi: 10.1016/j.apmr.2012.06.005. Epub 2012 Jun 18. PMID 22721868
- [Background] Katz-Leurer M, Rottem H, Meyer S. Hand-held dynamometry in children with traumatic brain injury: within-session reliability. Pediatr Phys Ther. 2008 Fall;20(3):259-63. doi: 10.1097/PEP.0b013e3181824782. PMID 18703964
- [Background] Ross SA, Engsberg JR. Relationships between spasticity, strength, gait, and the GMFM-66 in persons with spastic diplegia cerebral palsy. Arch Phys Med Rehabil. 2007 Sep;88(9):1114-20. doi: 10.1016/j.apmr.2007.06.011. PMID 17826455
- [Background] Engsberg JR, Ross SA, Collins DR. Increasing ankle strength to improve gait and function in children with cerebral palsy: a pilot study. Pediatr Phys Ther. 2006 Winter;18(4):266-75. doi: 10.1097/01.pep.0000233023.33383.2b. PMID 17108800
- [Background] Carey H, Martin K, Combs-Miller S, Heathcock JC. Reliability and Responsiveness of the Timed Up and Go Test in Children With Cerebral Palsy. Pediatr Phys Ther. 2016 winter;28(4):401-8. doi: 10.1097/PEP.0000000000000301. PMID 27661230
- [Background] Dewar R, Claus AP, Tucker K, Ware RS, Johnston LM. Reproducibility of the Kids-BESTest and the Kids-Mini-BESTest for Children With Cerebral Palsy. Arch Phys Med Rehabil. 2019 Apr;100(4):695-702. doi: 10.1016/j.apmr.2018.12.021. Epub 2019 Jan 9. PMID 30639271
- [Background] Badia M, Orgaz MB, Riquelme I, Gómez-Iruretagoyena J. Domains of the Cerebral Palsy Quality of Life Questionnaire (CP QOL) for Children and Adolescents: Spanish Adaptation and Psychometric Properties. 2021;33:331-349.
- [Result] Tinderholt Myrhaug H, Ostensjo S, Larun L, Odgaard-Jensen J, Jahnsen R. Intensive training of motor function and functional skills among young children with cerebral palsy: a systematic review and meta-analysis. BMC Pediatr. 2014 Dec 5;14:292. doi: 10.1186/s12887-014-0292-5. PMID 25475608
- [Result] Morgan C, Darrah J, Gordon AM, Harbourne R, Spittle A, Johnson R, Fetters L. Effectiveness of motor interventions in infants with cerebral palsy: a systematic review. Dev Med Child Neurol. 2016 Sep;58(9):900-9. doi: 10.1111/dmcn.13105. Epub 2016 Mar 29. PMID 27027732
- [Result] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Result] Ritzmann R, Stark C, Krause A. Vibration therapy in patients with cerebral palsy: a systematic review. Neuropsychiatr Dis Treat. 2018 Jun 18;14:1607-1625. doi: 10.2147/NDT.S152543. eCollection 2018. PMID 29950843
- [Result] Huang M, Liao LR, Pang MY. Effects of whole body vibration on muscle spasticity for people with central nervous system disorders: a systematic review. Clin Rehabil. 2017 Jan;31(1):23-33. doi: 10.1177/0269215515621117. Epub 2016 Jul 11. PMID 26658333
- [Result] Saquetto M, Carvalho V, Silva C, Conceicao C, Gomes-Neto M. The effects of whole body vibration on mobility and balance in children with cerebral palsy: a systematic review with meta-analysis. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):137-44. PMID 26032205
- [Result] Cheng HY, Yu YC, Wong AM, Tsai YS, Ju YY. Effects of an eight-week whole body vibration on lower extremity muscle tone and function in children with cerebral palsy. Res Dev Disabil. 2015 Mar;38:256-61. doi: 10.1016/j.ridd.2014.12.017. Epub 2015 Jan 7. PMID 25575288
- [Result] Cheng HY, Ju YY, Chen CL, Chuang LL, Cheng CH. Effects of whole body vibration on spasticity and lower extremity function in children with cerebral palsy. Hum Mov Sci. 2015 Feb;39:65-72. doi: 10.1016/j.humov.2014.11.003. Epub 2014 Nov 24. PMID 25461434
- [Result] Katusic A, Alimovic S, Mejaski-Bosnjak V. The effect of vibration therapy on spasticity and motor function in children with cerebral palsy: a randomized controlled trial. NeuroRehabilitation. 2013;32(1):1-8. doi: 10.3233/NRE-130817. PMID 23422453
- [Result] Park EY, Kim WH. Meta-analysis of the effect of strengthening interventions in individuals with cerebral palsy. Res Dev Disabil. 2014 Feb;35(2):239-49. doi: 10.1016/j.ridd.2013.10.021. Epub 2013 Nov 27. PMID 24291625
- [Result] Mockford M, Caulton JM. Systematic review of progressive strength training in children and adolescents with cerebral palsy who are ambulatory. Pediatr Phys Ther. 2008 Winter;20(4):318-33. doi: 10.1097/PEP.0b013e31818b7ccd. PMID 19011522
- [Result] Dodd KJ, Taylor NF, Graham HK. A randomized clinical trial of strength training in young people with cerebral palsy. Dev Med Child Neurol. 2003 Oct;45(10):652-7. doi: 10.1017/s0012162203001221. PMID 14515935
- [Result] Salem Y, Godwin EM. Effects of task-oriented training on mobility function in children with cerebral palsy. NeuroRehabilitation. 2009;24(4):307-13. doi: 10.3233/NRE-2009-0483. PMID 19597267
- [Result] Pandey, D. P., & Tyagi, V. (2011). Effect of functional strength training on functional motor performance in young children with cerebral palsy. Indian Journal of Physiotherapy and Occupational Therapy, 5(1), 52-55.
- [Result] Peungsuwan P, Parasin P, Siritaratiwat W, Prasertnu J, Yamauchi J. Effects of Combined Exercise Training on Functional Performance in Children With Cerebral Palsy: A Randomized-Controlled Study. Pediatr Phys Ther. 2017 Jan;29(1):39-46. doi: 10.1097/PEP.0000000000000338. PMID 27984466
- [Result] Gusso S, Munns CF, Colle P, Derraik JG, Biggs JB, Cutfield WS, Hofman PL. Effects of whole-body vibration training on physical function, bone and muscle mass in adolescents and young adults with cerebral palsy. Sci Rep. 2016 Mar 3;6:22518. doi: 10.1038/srep22518. PMID 26936535
- [Result] Pin TW, Butler PB, Purves S. Use of whole body vibration therapy in individuals with moderate severity of cerebral palsy- a feasibility study. BMC Neurol. 2019 May 1;19(1):80. doi: 10.1186/s12883-019-1307-5. PMID 31043157
- [Result] Taylor NF, Dodd KJ, Graham HK. Test-retest reliability of hand-held dynamometric strength testing in young people with cerebral palsy. Arch Phys Med Rehabil. 2004 Jan;85(1):77-80. doi: 10.1016/s0003-9993(03)00379-4. PMID 14970972